CLINICAL TRIAL: NCT03546712
Title: Standard References Norms for Tactile Localization Acuity in Upper Limb Among the Asymptomatic Middle School Children: A Normative Research
Brief Title: Estimating Error in Locating Touch Sensation on Forearm in Healthy Middle School Going Children
Status: Completed | Type: Observational
Sponsor: Maharishi Markendeswar University (Deemed to be University) (Other)
Responsible Party: Principal Investigator, Asir John Samuel, Associate professor of institute of physiotherapy and rehabilitation, Maharishi Markendeswar University (Deemed to be University)
Other Study IDs: MMDU/IEC/1188; U1111-1214-2489 (Other: UTN by WHO International Clinical Trial Registry)
Record Dates: First submitted 2018-05-23; First posted 2018-06-06 (Actual); Last update posted 2019-04-08 (Actual); Status verified 2019-04

CONDITIONS: Healthy
Keywords: Acuity; children; forearm; perception; touch location

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Tactile Localization — tactile localization is help to assess touch sensation

SUMMARY:
Tactile localization stimuli are fundamental in forearm to the somatosensory perception.Tactile localization reverse the touch internal organization of the forearm and in the normal development of children.It is helpful in quick estimation of tactile localization among the children in the age group, eight to thirteen years.Study design is cross-sectional study it is conducted from September 2017 to April 2019 and use stratified random sampling. subject recruitment is healthy school going children of age group between eight and thirteen year will be included in this study.The procedure will be explained to the children's before starting the test. Ascent will be obtained from the participant. Anthropometrics will be measured before beginning the procedure. The acuity of TL will be determined by the point-to-point tactile localization (PPTL) technique. For performing PPTL, the child will be seated and the examiner will locate a point on the participants forearm of the blinded child by a black pen marker. Then the child will be asked to relocate the point with the help of red pen marker in blindfolded state. The distance between black point and red point (in cm) will be noted this distance will be measure by measuring tape as the acuity of tactile localization. Mean of three readings will be used for estimating the normative reference value of tactile localization by PPTL technique.

DETAILED DESCRIPTION:
For performing Point to Point Tactile Localization, the child will be seated and the examiner will locate a point on the forearm of the blinded child by a black marker pen. Then the child will be asked to relocate the point with the help of red marked in blindfolded state. The distance between black point and red point (in cm) will be noted as the acuity of tactile localization. 15 areas in upper limb will be selected and PPTL will be performed on them. The fifteen areas are, phalanges of the palmer area of the little finger (palm 1), phalanx of the middle finger of the Palmer area (palm 2), phalanx of the thumb area of palm (palm 3), first dorsal interosseous (palm 4), mid last part of the forearm (forearm 1), middle of the medial forearm (forearm 2), medial side of the forearm (forearm 3), the lower portion of the arm (arm 1), middle posterior of arm (arm 2), lateral side of upper arm (arm 3), lower portion of medial arm (arm 4), middle portion of arm (arm 5), the median upper arm (arm 6), lower side arm (arm 7), and upper side of arm (arm 8). Mean of three readings will be used for estimating the normative reference value of tactile localization by PPTL technique.

ELIGIBILITY:
Inclusion Criteria: healthy school going children, Male and female, Age between eight-13 years, Able to understand commands, Obey simple comments

Exclusion Criteria: neurological diseases, disease of the skin, skin rashes, Non cooperative child, other medical conditions that prevent the from participating in the study

Ages: 8 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Healthy school going children age between eight and thirteen years without any neurological disease. healthy school children is able to follow commands and able to understand.
Sampling Method: Probability Sample
Enrollment: 365 (Actual)
Dates: Start 2018-11-12 (Actual); Primary Completion 2019-03-03 (Actual); Study Completion 2019-03-04 (Actual)

PRIMARY OUTCOMES:
distance in millimeter | 3 times
  distance between black pen marker and red pen marker point measure

CONTACTS AND LOCATIONS:
Overall Officials: Krati Omar, BPT, (MPT), Principal Investigator — Maharishi Markandeshwar Institute of physiotherapy and Rehabilitation
Locations (2):
- India (2):
  - Asir John Samuel, Ambāla, Haryana
  - Maharishi Markandeshwar Institute of physiotherapy and Rehabilitation, Ambāla, Haryana

IPD SHARING:
Plan to Share IPD: Undecided
undecided

REFERENCES:
- [Background] Pinto JM, Kern DW, Wroblewski KE, Chen RC, Schumm LP, McClintock MK. Sensory function: insights from Wave 2 of the National Social Life, Health, and Aging Project. J Gerontol B Psychol Sci Soc Sci. 2014 Nov;69 Suppl 2(Suppl 2):S144-53. doi: 10.1093/geronb/gbu102. PMID 25360015
- [Background] Ackerley R, Carlsson I, Wester H, Olausson H, Backlund Wasling H. Touch perceptions across skin sites: differences between sensitivity, direction discrimination and pleasantness. Front Behav Neurosci. 2014 Feb 19;8:54. doi: 10.3389/fnbeh.2014.00054. eCollection 2014. PMID 24600368
- [Background] Croy I, Sehlstedt I, Wasling HB, Ackerley R, Olausson H. Gentle touch perception: From early childhood to adolescence. Dev Cogn Neurosci. 2019 Feb;35:81-86. doi: 10.1016/j.dcn.2017.07.009. Epub 2017 Aug 18. PMID 28927641
- [Background] Rigato S, Banissy MJ, Romanska A, Thomas R, van Velzen J, Bremner AJ. Cortical signatures of vicarious tactile experience in four-month-old infants. Dev Cogn Neurosci. 2019 Feb;35:75-80. doi: 10.1016/j.dcn.2017.09.003. Epub 2017 Sep 14. PMID 28942240
- [Background] Harvie DS, Kelly J, Buckman H, Chan J, Sutherland G, Catley M, Novak J, Tuttle N, Sterling M. Tactile acuity testing at the neck: A comparison of methods. Musculoskelet Sci Pract. 2017 Dec;32:23-30. doi: 10.1016/j.msksp.2017.07.007. Epub 2017 Jul 29. PMID 28800436
- [Background] Chai G, Sui X, Li S, He L, Lan N. Characterization of evoked tactile sensation in forearm amputees with transcutaneous electrical nerve stimulation. J Neural Eng. 2015 Dec;12(6):066002. doi: 10.1088/1741-2560/12/6/066002. Epub 2015 Sep 24. PMID 26401550
- See also: Tactile acuity testing at the neck: A comparison of methods — https://doi.org/10.1016/j.msksp.2017.07.007